CLINICAL TRIAL: NCT03789760
Title: A Phase III, Randomised, Double-blind, Placebo-controlled, Parallel, and Multi-centre Study to Evaluate the Clinical Efficacy and Safety of SaiLuoTong (SLT) in the Treatment of Vascular Dementia
Brief Title: The Clinical Trial of Chinese Herbal Medicine (SaiLuoTong) Capsule
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shineway Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SW003
Record Dates: First submitted 2018-09-04; First posted 2018-12-31 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Vascular Dementia
Keywords: Vascular Dementia; cognitive
MeSH Terms: conditions — Dementia, Vascular | interventions — sailuotong

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active group (Experimental): take two pills (120 mg) of SaiLuoTong capsule each time, twice a day, 0.5 hours before breakfast and dinner, taking with lukewarm water.
  Interventions: Drug: SaiLuoTong capsule
- control group (Placebo Comparator): take two pills (120 mg) of placebo each time, twice a day, 0.5 hours before breakfast and dinner, taking with lukewarm water.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: SaiLuoTong capsule — 500 subjects are randomly divided into two groups by 3:1. 375 subjects in the active group take two pills(120mg) of SaiLuoTong capsule each time, twice a day, 0.5 hours before breakfast and dinner, taking with lukewarm water.
  Other Names: The effects of SaiLuoTong capsule on VaD
  Arms: active group
Drug: placebo — 500 subjects are randomly divided into two groups by 3:1. 125 subjects in the control group take two pills(120mg) of placebo each time, twice a day, 0.5 hours before breakfast and dinner, taking with lukewarm water.
  Arms: control group

SUMMARY:
As a traditional Chinese medicine compound, SaiLuoTong capsule is proven to have beneficial effects on learning and memory ability in animal models of vascular dementia (VaD). According to the result of the phase II study, the efficacy of SaiLuoTong capsule in the treatment of patients with VaD was better than that of placebo group and no difference in safety. So the study hypothesis is also that SaiLuoTong capsule will be effective in the treatment of patients with VaD and will be well tolerated. The purpose of the study is to confirm the efficacy and safety of SaiLuoTong capsule on patients with mild to moderate VaD. The outcome measures include general cognitive function, executive function, daily living skills, and mental behavior changes of symptoms in VaD patients.

DETAILED DESCRIPTION:
Vascular dementia (VaD) is a clinical syndrome of acquired intellectual and functional impairment that results from cerebrovascular diseases. SaiLuoTong capsule is a traditional Chinese medicine compound; it is composed of ginseng extract (the main composition: ginseng total saponins), ginkgo biloba extract (the main composition: YinXingTong ester) and safflower extract (the main composition: the west safflower total glycosides). The function of SaiLuoTong capsule is Yiqi Huoxue and Huayu Tongluo in Chinese traditional medicine theory. Pharmacodynamics studies showed that SaiLuoTong capsule can significantly improve neurological symptoms caused by focal cerebral ischemia in animals, and learning and memory ability in animal models of VaD. The result of the phase II study showed that the efficacy of SaiLuoTong capsule in the treatment of patients with VaD was better than that of placebo group and no difference in safety. Based on these previous evidences, the investigators conduct this study to further confirm the efficacy and safety of SaiLuoTong capsule in patients with mild to moderate VaD. This study is a phase III clinical trial of SaiLuoTong capsule for treatment of vascular dementia. The study is a 52-week, multicentre, randomized, double -blind, placebo-controlled study.

ELIGIBILITY:
Inclusion Criteria:

* 40 years≤Age≤75 years, female or male.
* With an education at more than (including) 6 years.
* Meet the diagnostic criteria for dementia in Diagnostic and Statistical Manual of Mental Disorders-5th Edition (DSM-V).
* Meet the National Institute of Neurological Disorders and Stroke-Association Internationale pour la Recherche etl'Enseignement en Neurosciences(NINDS-AIREN) Criteria of Probable Vascular Dementia (1993).
* MRI (magnetic resonance imaging) supports the presence of ischemic cerebrovascular disease, and meets NINDS-AIREN Imaging Criteria; the diameter of each infarct≤ 30mm(And the perivascular spaces and cerebral microbleeds were excluded).
* Modified Hachinski Ischemic (mHIS) Scale ≥ 4.
* Hamilton depression scale (HAMD) ≤ 17.
* Patients with mild or moderate VaD: 10 ≤ MMSE ≤ 26 and 1 ≤ CDR ≤ 2.
* Willing to participate in this study and could sign the informed consent form by him/herself and lawful guardian prior to the study.
* The subjects must have a care giver who are cognitively normal (MMSE scores: illiteracy> 17 points, 1 - 6 years of education > 20 points, 7 years and above of education > 24 points). The care giver shall also be able to take care of the patient at least 4 days a week for more than 4 hours a day while he or she can accompany the subjects to attend each visit. During the trial, a new caregiver must have MMSE score and the results would be presented in forms of subjects in the attachment.

Exclusion Criteria:

* Patients with dementia caused by a brain disease other than VaD (such as Alzheimer's disease, dementia with Lewy bodies, frontotemporal dementia, Parkinson's disease, central nervous system demyelinative diseases, tumour, hydrocephalus, trauma, central nervous system infection, such as syphilis, AIDS and Creutzfeldt-Jakob disease);
* Patients with serious neurological impairment to finish the examination: hand hemiplegia, aphasia, and visual or hearing impairment.
* Laboratory anomalies: hemoglobin (Hb) level less than 80g/L , platelet count (Plt) level less than 50×109/L, activated partial thromboplastin time (APTT) exceeds 2.5 times the normal upper level, fibrinogen(FIB) level less than 0.5g/L, prothrombin time (PT) exceeds 2.5 times the normal upper level, Serum creatinine (Scr) exceeds 3 times the normal upper level, alanine aminotransferase (ALT) exceed 5 times the normal upper level , aspartate aminotransferase (AST) exceed 5 times the normal upper level, alkaline phosphates (ALP) exceed 5 times the normal upper level , γ-glutamyl transferase (γ-GT) exceed 5 times the normal upper level, total bilirubin (TBiL) exceeds 3 times the normal upper level.
* The subjects have nutritional and metabolic diseases and endocrine system diseases that cannot been controlled by therapy - thyroid diseases, parathyroid disease, vitamin or element deficiency.
* Patients with serious circulatory system diseases, respiratory system diseases, urinary system diseases, digestive system diseases, haemopoietic system diseases (such as unstable angina, uncontrollable asthma and active gastrorrhagia) and cancer.
* Serious mental disease (such as depression and schizophrenia) and epilepsy.
* Gastrointestinal diseases that may affect the absorption, distribution, and metabolism of the investigational drug.
* Alcohol and drug abuse.
* Patients who have been given any drug that can affect the cognitive function (including Chinese herbal preparations containing any one of these: ginseng, ginkgo leaf, and saffron; Western medicines such as donepezil, karbalatine, rivastigmine, huperzine a, memantine and similar drugs, etc; Butylphthalide and other drugs with the same effect such as runeirergine, aniracetam, cytosporine, dihydroergine, nimodipine, etc) within one month before the start of this study and cannot be discontinued.
* Patients who are allergic to more than 2 drugs or any component of the SLT capsules.
* Pregnant or lactating women.
* Patients who have participated in other clinical studies within 3 months prior to this study.
* Cannot accept magnetic resonance imaging (MRI) examination.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 493 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-05-19 (Actual)

PRIMARY OUTCOMES:
Vascular Dementia Assessment Scale-cognitive Subscale(VaDAS-cog) | Change from baseline VaDAS-cog score at Week 52
  The VaDAS-cog comprises the Alzheimer's disease assessment scale(ADAS-cog) plus the Maze and Number Cancellation test to specifically assess executive function. The score of each item is summed to compute a total score. The range of the total score was from 0(no cognitive impairment) to 90(severe cognitive impairment). The data in the table below is the statistical data (mean,SD) of precise scores at screening and week 0 (baseline), while the statistical data of difference value compared to the score of Baseline at weeks 52.
Alzheimer's Disease Cooperative Study-clinical Global Impression of Change(ADCS-CGIC) | Change from baseline ADCS-CGIC score at Week 52
  The Alzheimer's Disease Cooperative Study-clinical Global Impression of Change(ADCS-CGIC) involves comparison of data acquisition from both home and clinic and the use of both informant-ratings and self-ratings. Important outcomes include clinical global impressions of change (CGIC) as indicators of clinically meaningful change. In week 0 (baseline), the score was to judge the severity of the cognitive, 0(no evaluate),1(normal),2(slight intelligence obstacle),3(mide intelligence obstacle),4(moderate intelligence obstacle),5(significantly intelligence obstacle),6(severe intelligence obstacle),7(intelligent obstacle end-stage). In week 13,26,39,52, the score was to judge the change of the clinical global impression,1(improved significantly),2(improve),3(improve a little),4(no change),5(a little deteriorated),6(deteriorated),7(serious deterioration).

SECONDARY OUTCOMES:
Alzheimer's Disease Cooperative Study-activities of Daily Living(ADCS-ADL) | Change from baseline ADCS-ADL score at Week 26
  To assess the daily living activity of the patients, including a subgroup in which there are 23 items to be checked and the total score is 78. A higher score represents a better daily living activity, vice versa. The score of each item is summed to compute a total score. The data in the table below is the statistical data (mean,SD) of precise scores at week 0 (baseline), while the statistical data of difference value compared to the score of baseline at weeks 26.
Alzheimer's Disease Cooperative Study-activities of Daily Living(ADCS-ADL) | Change from baseline ADCS-ADL score at Week 52
  To assess the daily living activity of the patients, including a subgroup in which there are 23 items to be checked and the total score is 78. A higher score represents a better daily living activity, vice versa. The score of each item is summed to compute a total score. The data in the table below is the statistical data (mean,SD) of precise scores at week 0 (baseline), while the statistical data of difference value compared to the score of baseline at weeks 52.
Mini-mental State Examination(MMSE) | Change from baseline MMSE score at Week 26
  The MMSE is a global test of cognitive function, for which the total score ranges from 0 to 30, with higher scores indicating lesser severity. The score of each item is summed to compute a total score. The data in the table below is the statistical data (mean, SD) of precise scores at screening (baseline), while the statistical data of difference value compared to the score of baseline at weeks 26.
Mini-mental State Examination(MMSE) | Change from baseline MMSE score at Week 52
  The MMSE is a global test of cognitive function, for which the total score ranges from 0 to 30, with higher scores indicating lesser severity. The score of each item is summed to compute a total score. The data in the table below is the statistical data (mean, SD) of precise scores at screening (baseline), while the statistical data of difference value compared to the score of baseline at weeks 52.
Clinical Dementia Rating(CDR Scale ) | Change from baseline CDR Scale score at Week 26
  The CDR is a numeric scale used to quantify the severity of symptoms of dementia (i.e. its 'stage'). Talk to the patients or those who know well about the patients and assess the 6 functions (memory, orientation, judgment and problem-solving ability, social activities, household duties and hobbies as well as self-care ability) to obtain the scores and based on the predetermined principles the CDR score is calculated. The diagnostic criteria[68]: normal-CDR=0; suspected dementia-CDR=0.5, mild dementia-CDR=1; moderate dementia- CDR=2; and serious dementia-CDR=3. The data in the table below is the statistical data (mean, SD) of precise scores at baseline and weeks 26.
Clinical Dementia Rating(CDR Scale ) | Change from baseline CDR Scale score at Week 52
  The CDR is a numeric scale used to quantify the severity of symptoms of dementia (i.e. its 'stage'). Talk to the patients or those who know well about the patients and assess the 6 functions (memory, orientation, judgment and problem-solving ability, social activities, household duties and hobbies as well as self-care ability) to obtain the scores and based on the predetermined principles the CDR score is calculated. The diagnostic criteria[68]: normal-CDR=0; suspected dementia-CDR=0.5, mild dementia-CDR=1; moderate dementia- CDR=2; and serious dementia-CDR=3. The data in the table below is the statistical data (mean, SD) of precise scores at baseline and weeks 52.
Clinical Dementia Rating sum of boxes(CDR-sb) | Change from baseline CDR-sb score at Week 26
  CDR-sb is the sum of boxes of CDR, with higher scores indicating severer degree of impairment. CDR-sb is the algebraic sum of 6 functional domains with a range of 0(normal) - 18(severe dementia). The data in the table below is the statistical data (mean,SD) of precise scores at weeks 0 (baseline), while the statistical data of difference value compared to the score of baseline at weeks 26.
Clinical Dementia Rating sum of boxes(CDR-sb) | Change from baseline CDR-sb score at Week 52
  CDR-sb is the sum of boxes of CDR, with higher scores indicating severer degree of impairment. CDR-sb is the algebraic sum of 6 functional domains with a range of 0(normal) - 18(severe dementia). The data in the table below is the statistical data (mean,SD) of precise scores at weeks 0 (baseline), while the statistical data of difference value compared to the score of baseline at weeks 52.
Blood biomarker: Brain-derived neurotrophic factor(BDNF) | Change from baseline BDNF at Week 26
  The data in the table below is the statistical data (mean,SD) of precise measurement at weeks 0 (baseline), while the statistical data of difference value compared to the score of baseline at weeks 26.
Blood biomarker: Brain-derived neurotrophic factor(BDNF) | Change from baseline BDNF at Week 52
  The data in the table below is the statistical data (mean,SD) of precise measurement at weeks 0(baseline), while the statistical data of difference value compared to the score of baseline at weeks 52.
Blood biomarker: Vascular endothelial growth factor(VEGF) | Change from baseline VEGF at Week 26
  The data in the table below is the statistical data (mean,SD) of precise measurement at weeks 0 (baseline), while the statistical data of difference value compared to the score of baseline at weeks 26.
Blood biomarker: Vascular endothelial growth factor(VEGF) | Change from baseline VEGF at Week 52
  The data in the table below is the statistical data (mean,SD) of precise measurement at weeks 0 (baseline), while the statistical data of difference value compared to the score of baseline at weeks 52.
Blood biomarker: Matrix metalloproteinase-9(MMP-9) | Change from baseline MMP-9 at Week 26
  The data in the table below is the statistical data (mean,SD) of precise measurement at weeks 0 (baseline), while the statistical data of difference value compared to the score of baseline at weeks 26.
Blood biomarker: Matrix metalloproteinase-9(MMP-9)) | Change from baseline MMP-9 at Week 52
  The data in the table below is the statistical data (mean,SD) of precise measurement at weeks 0 (baseline), while the statistical data of difference value compared to the score of baseline at weeks 52.
Blood biomarker: Interleukin-6(IL-6) | Change from baseline MMP-9 at Week 26
  The data in the table below is the statistical data (mean,SD) of precise measurement at weeks 0 (baseline), while the statistical data of difference value compared to the score of baseline at weeks 26.
Blood biomarker: Interleukin-6(IL-6) | Change from baseline MMP-9 at Week 52
  The data in the table below is the statistical data (mean,SD) of precise measurement at weeks 0 (baseline), while the statistical data of difference value compared to the score of baseline at weeks 52.
Vascular Dementia Assessment Scale-cognitive Subscale(VaDAS-cog) | Change from baseline VaDAS-cog score at week 13
  The VaDAS-cog comprises the ADAS-cog plus the Maze and Number Cancellation test to specifically assess executive function. The score of each item is summed to compute a total score. The range of the total score was from 0(no cognitive impairment) to 90(severe cognitive impairment). The data in the table below is the statistical data (mean,SD) of precise scores at screening and week 0 (baseline), while the statistical data of difference value compared to the score of Baseline at weeks 13.
Vascular Dementia Assessment Scale-cognitive Subscale(VaDAS-cog) | Change from baseline VaDAS-cog score at week 26
  The VaDAS-cog comprises the ADAS-cog plus the Maze and Number Cancellation test to specifically assess executive function. The score of each item is summed to compute a total score. The range of the total score was from 0(no cognitive impairment) to 90(severe cognitive impairment). The data in the table below is the statistical data (mean,SD) of precise scores at screening and week 0 (baseline), while the statistical data of difference value compared to the score of Baseline at weeks 26.
Vascular Dementia Assessment Scale-cognitive Subscale(VaDAS-cog) | Change from baseline VaDAS-cog score at week 39
  The VaDAS-cog comprises the ADAS-cog plus the Maze and Number Cancellation test to specifically assess executive function. The score of each item is summed to compute a total score. The range of the total score was from 0(no cognitive impairment) to 90(severe cognitive impairment). The data in the table below is the statistical data (mean,SD) of precise scores at screening and week 0 (baseline), while the statistical data of difference value compared to the score of Baseline at weeks 39.
Alzheimer's Disease Cooperative Study-clinical Global Impression of Change(ADCS-CGIC) | Change from baseline ADCS-CGIC score at week 13
  The ADCS-CGIC involves comparison of data acquisition from both home and clinic and the use of both informant-ratings and self-ratings. Important outcomes include clinical global impressions of change (CGIC) as indicators of clinically meaningful change. In week 0 (baseline), the score was to judge the severity of the cognitive, 0(no evaluate),1(normal),2(slight intelligence obstacle),3(mide intelligence obstacle),4(moderate intelligence obstacle),5(significantly intelligence obstacle),6(severe intelligence obstacle),7(intelligent obstacle end-stage). In week 13,26,39,52, the score was to judge the change of the clinical global impression,1(improved significantly),2(improve),3(improve a little),4(no change),5(a little deteriorated),6(deteriorated),7(serious deterioration).
Alzheimer's Disease Cooperative Study-clinical Global Impression of Change(ADCS-CGIC) | Change from baseline ADCS-CGIC score at week 26
  The ADCS-CGIC involves comparison of data acquisition from both home and clinic and the use of both informant-ratings and self-ratings. Important outcomes include clinical global impressions of change (CGIC) as indicators of clinically meaningful change. In week 0 (baseline), the score was to judge the severity of the cognitive, 0(no evaluate),1(normal),2(slight intelligence obstacle),3(mide intelligence obstacle),4(moderate intelligence obstacle),5(significantly intelligence obstacle),6(severe intelligence obstacle),7(intelligent obstacle end-stage). In week 13,26,39,52, the score was to judge the change of the clinical global impression,1(improved significantly),2(improve),3(improve a little),4(no change),5(a little deteriorated),6(deteriorated),7(serious deterioration).
Alzheimer's Disease Cooperative Study-clinical Global Impression of Change(ADCS-CGIC) | Change from baseline ADCS-CGIC score at week 39
  The ADCS-CGIC involves comparison of data acquisition from both home and clinic and the use of both informant-ratings and self-ratings. Important outcomes include clinical global impressions of change (CGIC) as indicators of clinically meaningful change. In week 0 (baseline), the score was to judge the severity of the cognitive, 0(no evaluate),1(normal),2(slight intelligence obstacle),3(mide intelligence obstacle),4(moderate intelligence obstacle),5(significantly intelligence obstacle),6(severe intelligence obstacle),7(intelligent obstacle end-stage). In week 13,26,39,52, the score was to judge the change of the clinical global impression,1(improved significantly),2(improve),3(improve a little),4(no change),5(a little deteriorated),6(deteriorated),7(serious deterioration).

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Jia, Professor, Principal Investigator — Xuan Wu Hospital of Capital Medical University
Locations (29):
- China (29):
  - Xuan Wu Hospital of Capital Medical University, Beijing, Beijing Municipality
  - Peking University Shougang Hospital, Beijing, Beijing Municipality
  - Xiyuan Hospital, Beijing, Beijing Municipality
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Affiliated Hospital of Chengde Medical College, Chengde, Hebei
  - Handan First Hospital, Handan, Hebei
  - Hebei Central Hospital of petrochina, Langfang, Hebei
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Fourth Hospital of Medical University, Harbin, Hei Longjiang
  - The First People's Hospital of Luoyang, Luoyang, Henan
  - The First affiliated Hospital of Nanyang Medical college, Nanyang, Henan
  - Nanyang Second People's Hospital, Nanyang, Henan
  - The First Hospital of Changsha, Changsha, Hunan
  - Xiangya Boai Rehability Hospital, Changsha, Hunan
  - Yueyang Second People's Hospital, Yueyang, Hunan
  - Baogang Hospital, Baotou, Inner Mongolia
  - Inner Mongolia International Mongolian Hospital, Hohhot, Inner Mongolia
  - Taizhou Hospital of Chinese Medicine, Taizhou, Jiangsu
  - Jiujiang University Clinical Medical College ▪ Jiujiang University Hospital, Jiujiang, Jiangxi
  - Nanchang Hongdu Hospital of TCM, Nanchang, Jiangxi
  - Changzhi People's Hospital, Changzhi, Shanxi
  - Jinzhong First People's Hospital, Jinzhong, Shanxi
  - Xianyang Hospital of Yan'an University, Xianyang, Shanxi
  - Yuncheng Central Hospital, Yuncheng, Shanxi
  - The Second people's Hospital of Neijiang, Neijiang, Sichuan
  - Second Teaching Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality
  - The Second Hospital of Xingjiang Medical University, Ürümqi, Xingjiang
  - The Central Hospital of Lishui City, Lishui, Zhejiang